CLINICAL TRIAL: NCT00256568
Title: Outpatient Prescription Errors: Detection, Analysis, and Impact on Safety
Status: Completed | Type: Observational
Sponsor: University of Vermont (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Vermont Program for Quality in Health Care (Other)
Responsible Party: Principal Investigator, Amanda Kennedy, Assistant Professor of Medicine, University of Vermont
Other Study IDs: K08HS013891 (AHRQ)
Record Dates: First submitted 2005-11-17; First posted 2005-11-21 (Estimated); Last update posted 2011-12-15 (Estimated); Status verified 2011-12

CONDITIONS: Medication Errors
Keywords: Medical Errors; Medication Errors; Prescriptions, Drug; Pharmacies; Ambulatory Care Facilities
MeSH Terms: interventions — Adverse Drug Reaction Reporting Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Primary Care Practices: One hundred and three prescribers, managers, nurses and office staff at seven primary care practices in Vermont
  Interventions: Behavioral: reporting system

INTERVENTIONS:
Behavioral: reporting system — Nurses and office staff were asked to report all communications with community pharmacists regarding prescription problems

SUMMARY:
The purpose of this study is to better understand outpatient prescribing errors through clinic and pharmacy-based error reporting systems.

DETAILED DESCRIPTION:
Medication errors cause substantial morbidity and mortality in the United States. However, relatively little is known about medication errors in the outpatient setting. The broad goal of this proposal is to improve outpatient safety. Specifically, this research plan promotes the understanding of the causes of outpatient prescription errors. The specific aims of this project are:

1. To develop and evaluate a novel reporting system in physicians' offices for detecting prescription errors
2. To develop and evaluate a novel improvement system in community pharmacies to increase prescription error reporting by pharmacists
3. To analyze reports of outpatient prescription errors and understand their root causes

To achieve these specific aims, statewide research will be conducted utilizing qualitative and quantitative methods including root cause analysis, failure mode and effects analysis, and surveys. This research plan will promote patient safety by furthering the understanding of the causes of outpatient prescription errors in all outpatient populations, including rural, women, children, elderly, low income, and the chronically ill.

ELIGIBILITY:
Inclusion Criteria:

* Employed in a physician's office or community pharmacy

Exclusion Criteria:

* Not employed in a physician's office or community pharmacy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary Care Practices
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2003-09; Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda G Kennedy, PharmD, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont, Division of General Internal Medicine, Burlington, Vermont, United States

REFERENCES:
- [Background] Kennedy AG, Littenberg B. Medication error reporting by community pharmacists in Vermont. J Am Pharm Assoc (2003). 2004 Jul-Aug;44(4):434-8. doi: 10.1331/1544345041475724. PMID 15372863
- [Background] Kennedy AG, Littenberg B, Vezina LC. Vioxx-Viagra confusion. Am J Health Syst Pharm. 2002 Nov 1;59(21):2112. doi: 10.1093/ajhp/59.21.2112a. No abstract available. PMID 12434730
- [Result] Kennedy AG, Littenberg B, Senders JW. Using nurses and office staff to report prescribing errors in primary care. Int J Qual Health Care. 2008 Aug;20(4):238-45. doi: 10.1093/intqhc/mzn015. Epub 2008 Apr 22. PMID 18430748